CLINICAL TRIAL: NCT05920343
Title: Prevention of Thromboembolism With Rivaroxaban in Genitourinary Cancer Patients Receiving Systemic Therapy: A Randomized Placebo-Controlled, Double-Blind Clinical Trial
Brief Title: VTE Prevention With Rivaroxaban in Genitourinary Cancer Patients Receiving Systemic Therapy
Acronym: PREVENT-GU
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network); Kidney Cancer Research Network of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PGU2023
Record Dates: First submitted 2023-06-08; First posted 2023-06-27 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Venous Thromboembolism; Urologic Cancer
Keywords: Genitourinary Cancer; Venous Thromboembolism; Systemic Therapy; Thromboprophylaxis
MeSH Terms: conditions — Venous Thromboembolism; Urologic Neoplasms; Urogenital Neoplasms | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Participants receiving study drug (Rivaroxaban)
  Interventions: Drug: Rivaroxaban 10 MG
- Control (Placebo Comparator): Participants receiving matched placebo
  Interventions: Other: Placebo control

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — The intervention in the experimental arm will be rivaroxaban, 10 mg PO once daily (prophylactic dosing) for 180 days after the start of systemic therapy or until one of the primary study outcomes occurs (VTE or major bleeding).
  Other Names: Xarelto
  Arms: Rivaroxaban
Other: Placebo control — Identical to Rivaroxaban intervention except participants will receive a matched placebo instead of the study drug
  Arms: Control

SUMMARY:
Patients with genitourinary cancers (ex: bladder, testicular, kidney) are at high risk of developing blood clots if they receive systemic therapy (ex: chemotherapy, immunotherapy). Blood clots cause pain, may require hospitalization and invasive testing, and in some cases cause death. In fact, blood clots are one of the leading causes of death in patients with cancer. Furthermore, patients who develop a blood clot require medication to thin the blood for a prolonged (sometimes indefinite) period of time, and this can disrupt other important cancer treatments. Studies have shown that using low dose blood thinners to prevent blood clots during systemic therapy is effective in some patients with cancer. However very few patients in these studies had genitourinary cancers, therefore physicians in Canada are not sure if recommending blood thinners to patients with genitourinary cancers is useful or safe. Safety is a primary concern because blood thinners may cause bleeding, and patients with genitourinary cancers may have higher risk of bleeding than patients with other types of cancer. The investigators hypothesize that blood thinners are effective and safe for reducing blood clots in patients with genitourinary cancers. The objective of this study is to determine if a large clinical trial testing the effectiveness and safety of low dose blood thinners for preventing blood clots in patients with genitourinary cancers receiving systemic therapy is feasible.

DETAILED DESCRIPTION:
Background and Importance: Patients with cancer receiving systemic therapy are at high risk of venous thromboembolism (VTE). Thromboprophylaxis with antiocoagulants reduces VTEs during chemotherapy by 60%. Despite this, thromboprophylaxis is not routinely used in Canada for patients with genitourinary (GU) malignancies (bladder, testis, kidney). Reasons prophylaxis is not used are that very few GU patients were included in landmark trials evaluating DOACs, and because GU patients may be at higher risk of bleeding compared to non-GU cancer patients. The omission of GU patients from prior trials has created an important gap in knowledge because these patients have among the highest risk of VTE of all cancer patients. Prior studies have reported VTE rates during chemotherapy for bladder and testis cancer in the range of 10-15%, well above thresholds at which guidelines usually recommend thromboprophylaxis.

Hypotheses: The investigators hypothesize that thromboprophylaxis with a direct oral anticoagulant (DOAC) during systemic therapy for GU malignancies will reduce the risk of VTE with acceptable risk of major bleeding. Secondly, the investigators hypothesize that a randomized trial of thromboprophylaxis versus placebo in GU patients is feasible and needed to change care in Canada.

Research goals: The goal of this pilot study is to determine if a randomized control trial of thromboprophylaxis with rivaroxaban versus placebo in GU patients receiving systemic therapy is feasible.

Methods: This internal pilot feasibility study will randomize patients with GU malignancies receiving systemic therapy (patients) to rivaroxaban 10mg daily (intervention) versus placebo (control). The primary outcome of this internal pilot study will be feasibility of patient accrual. Feasibility will be reported as the average number of patients enrolled per month. Secondary outcomes will be time to trial initiation, number of patients enrolled per site, and proportion of patients who complete the intervention. If feasibility is confirmed, patients enrolled in the pilot will be included in the full trial using a vanguard design.

The primary outcome(s) of the full trial will be VTE (efficacy outcome) and major bleeding (safety outcome) during the intervention. Patient reported outcomes including quality of life will also be recorded.

Expected outcomes: While thromboprophylaxis is effective in cancer patients, medical guidelines only recommend prophylaxis for some patients due to limited evidence in disease-specific subgroups. Importantly, safety concerns in GU patients are a particular concern necessitating further study of this population. The investigators expect the results of this internal pilot study to prove feasibility of a full trial. The full trial will determine the net benefits/harms of prophylaxis in GU patients and change practice worldwide, regardless of the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are starting systemic therapy for active GU cancer (bladder, testis, ureter/renal pelvis, kidney, urethral, penile) except for prostate cancer.
* Age ≥ 18
* Eligible systemic therapies include chemotherapy, targeted therapies (tyrosine kinase inhibitors and antiangiogenic therapy), and immunotherapies.
* Patients must be initiating systemic therapy with a minimum planned treatment duration of 8 weeks.

Exclusion Criteria:

* Anticoagulation (prophylactic or therapeutic dosing) required for another indication for entire duration of study
* Known allergies to rivaroxaban
* Concomitant use of dual antiplatelet therapy (two antiplatelet medications oncomitantly)
* Ongoing refractory bleeding that may be exacerbated by rivaroxaban.
* Concomitant use of strong inducers or inhibitors of CYP3A4 or glycoprotein-P (known interaction with rivaroxaban).
* Severe renal insufficiency (Creatinine clearance <30 mL/min (defined by Cockcroft-Gault))
* Severe liver disease (e.g. acute clinical hepatitis, chronic active hepatitis, cirrhosis)
* Thrombocytopenia < 50 x 109/L
* Life expectancy under 6 months.
* Pregnancy (if child bearing age under 50 and sexually active, documentation of use of effective contraception or negative B- HCG is required)
* Patient is breastfeeding or lactating
* History of condition at increased bleeding risk including, but not limited to:

cerebral infarction (hemorrhagic or ischemic), active peptic ulcer disease with recent bleeding, spontaneous or acquired impairment of hemostasis in the previous 4 weeks.

* Chronic hemorrhagic disorder
* Inability to adhere to protocol or obtain consent.
* Patients may be excluded from the study for other reasons, at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment, assesed by the number of patients accrued per month | Enrollment
  The primary outcome of this Pilot Trial is feasibility of enrollment. Feasibility will be measured by the average number of patients accrued per month.

SECONDARY OUTCOMES:
Adherence to the study intervention, assessed as the proportion of patients taking the study medication >80% of days taken during the study period, | During 180 days of study intervention
  This outcome will measure patient adherence to the study intervention (defined as >80% of medication taken during the study intervention period). This will be assessed using pill counts during study follow-ups.
Recruitment rate | Enrollment
  Number of participants recruited per month at each study site
VTE incidence | During 180 days of study intervention
  VTE will be recorded and adjudicated similarly to the full trial. Outcomes will be examined in aggregate to ascertain an estimate of baseline risk for patients in the trial. VTE outcomes will NOT be examined or reported by allocation group in the Pilot so all patients can be included in Full Trial analyses (internal pilot design).
Bleeding incidence | During 180 days of study intervention
  Bleeding outcomes (major and minor) will be recorded and adjudicated similarly to the full trial. Outcomes will be examined in aggregate to ascertain an estimate of baseline risk for patients in the trial. Bleeding outcomes will NOT be examined or reported by allocation group in the Pilot so all patients can be included in Full Trial analyses (internal pilot design).

OTHER OUTCOMES:
VTE-related death | During 180 days of study intervention
  VTE-related death will be collected during the pilot but will not be analyzed until the full trial. VTE-related death will assess the frequency of deaths among participants directly related to a VTE event.
Overall survival | During 180 days of study intervention
  Overall survival will be collected during the pilot but will not be analyzed until the full trial. Overall survival will assess the frequency with which participants die by any cause during the intervention.
Health-related Quality of Life assessed using the EQ-5D-5L Score | During 180 days of study intervention
  Health-related Quality of Life will be collected during the pilot but will not be analyzed until the full trial. Health-related Quality of Life will be assessed using the EQ-5D-5L questionnaire. EQ-5D-5L contains two scores: The VAS ranges from 0-100 and represents a patient's sense of their overall health. Higher VAS scores represent a better outcome. The second measure is the EQ-5D-5L index which ranges from 0-1 (scores are reported with three decimal points) and shows quality of life along 5 dimensions which are weighted based on regional values in the final index score. Higher index scores represent a better outcome
Incremental cost-effectiveness ratio | During 180 days of study intervention
  Incremental cost-effectiveness ratio will be collected during the pilot but will not be analyzed until the full trial. Incremental cost-effectiveness ratio will take the form of a cost utility analysis with outcome expressed as incremental cost per quality adjusted life year (QALY) gained.

CONTACTS AND LOCATIONS:
Overall Officials: Luke T Lavallee, MDCM MSc FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers.